CLINICAL TRIAL: NCT06860828
Title: Risk and Resilience, Clinical Presentation, and Biomarker Profiles of Chronic Traumatic Encephalopathy and Related Dementias: The DIAGNOSE CTE Research Project-II
Brief Title: The DIAGNOSE CTE Research Project-II
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of California, San Francisco (UCSF) Alzheimer Disease Research Center (ADRC) (Unknown); 1Florida ADRC, University of Florida (Unknown); University of Texas Health Science Center at San Antonio (South Texas) ADRC (Unknown); Laboratory of Neuro Imaging (LONI) at University of Southern California (USC) (Unknown); Concussion Legacy Foundation (CLF) (Unknown); Banner Alzheimer's Institute (Other)
Responsible Party: Sponsor
Other Study IDs: H-45461; 1R01NS139383-01 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-03-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Traumatic Encephalopathy (CTE); Alzheimer Disease; Alzheimer Disease and Related Dementias (ADRD); Brain Injuries, Traumatic
Keywords: Traumatic encephalopathy syndrome (TES); Repetitive head impacts (RHI); Former national football league players; Former varsity level college football players; Neuroimaging
MeSH Terms: conditions — Chronic Traumatic Encephalopathy; Alzheimer Disease; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from the buffy coat for APOE genotyping as well as to develop a genetic risk score algorithm for CTE. Interactions between RHI and select Single Nucleotide Polymorphisms (SNPs) will be used to examine the modification of RHI-related risk by genetic susceptibility for CTE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Former college and professional football players: 150 football players from DIAGNOSE I and an additional 75 former college and football players will be enrolled in DIAGNOSE II for a total anticipated cohort size of 225.
- Asymptomatic non-RHI/Controls: 50/60 controls from DIAGNOSE I and an additional 25 controls will be enrolled in DIAGNOSE II for a total anticipated cohort size of 75.
- Cognitive impairment due to Alzheimer's disease (AD-CI): 50 participants with cognitive impairment due to AD will be enrolled in DIAGNOSE II for an anticipated cohort size of 50.

SUMMARY:
Each year, millions of people are exposed to repetitive head impacts (RHI) through contact sports. RHI can result in concussions and asymptomatic non-concussions to confer risk for Alzheimer's disease (AD) and related dementias (ADRD) including chronic traumatic encephalopathy (CTE). Presently, a diagnosis of CTE can only be rendered at autopsy and it has been neuropathological diagnosed in several hundreds of American football players particularly those who played at elite levels (college and professional). The ability to make an accurate diagnosis of CTE is needed to facilitate research on risk factors, mechanisms, prevention, and treatment.

In 2015, the investigators were awarded a NINDS funded 7-year U01 known as the DIAGNOSE CTE Research Project (NCT02798185) designed to develop biomarkers, characterize the clinical presentation, and examine genetic and RHI risk factors for CTE. This current 5-year NIH funded multicenter study DIAGNOSE CTE Research Project-II will build on and extend those findings.

DETAILED DESCRIPTION:
The aims of the DIAGNOSE CTE Research Project-II are to:

* retain and grow DIAGNOSE-I and examine the clinical and biomarker course of Traumatic Encephalopathy Syndrome (TES);
* investigate risk and resilience factors of TES; and
* compare biomarkers of amyloid (Aβ), p-tau, neurodegeneration, neuroinflammation, and white matter (WM) injury between TES and AD.

The investigators hypothesize that TES has unique clinical and biomarker profiles, and RHI and non-RHI risk factors influence the development of TES.

There will be 3 study groups:

1. Retention, 150 former football players and 50 controls retained from DIAGNOSE-I;
2. Expansion, the investigators will grow DIAGNOSE-I by newly recruiting 75 former college and professional football players and 25 controls;
3. AD, 50 Aβ+ participants with cognitive impairment. In total, the investigators will study 225 former football players, 75 controls, and 50 AD.

Participants will complete a single visit, including clinical exams, social determinants of health (SDOH) measures, MRI, blood draw, and tau PET, at 1 of 5 P30 AD Research Centers (ADRCs): Boston University (BU), University of California, San Francisco (UCSF), Arizona/Banner Alzheimer's Institute (BAI), University of Florida (1Florida), and University of Texas Health Science Center at San Antonio (South Texas).

The Retention Cohort will have 18F-Flortaucipir (18F-AV-1451, Tauvid (FTP)) PET to study its longitudinal value. The Expansion Cohort will have 18F-MK-6240 (MK-6240) PET to build on the investigators' preliminary data. A subset of the Retention Cohort (n=20) will have FTP and MK-6240 for tracer comparison. Blood will be analyzed for 6 p-tau epitopes, Aβ40/42, neuroinflammation, and WM injury. DIAGNOSE-I participants were asked to pledge to donate their brain.

This study will permit continued brain donation and clinical-pathological validation studies. Results will provide insight into the detection, diagnosis, and prognosis for people living with CTE, paving the way for treatment trials.

ELIGIBILITY:
Inclusion Criteria:

1. Former college or professional football players (n=225) will include those retained from DIAGNOSE-I (n=150) and newly recruited (n=75). Criteria will include

   1. Former college football players must have played more than 6 years of football including 3 or more years at the college level. They must not have played organized football or other contact sports following college.
   2. Former professional football players must have played 12 or more years of total football including 3 or more years in college and 4 or more seasons professionally.
2. Control (n=75) will include those retained from DIAGNOSE-I (n=50) and newly recruited (n=25). Inclusion criteria for control include:

   1. Asymptomatic at screening
   2. Never been diagnosed with, or treated for, any of the following: depression, manic-depressive or bipolar disorder, anxiety, or other psychiatric or mental health problems
   3. No known traumatic brain injury (TBI) and/or moderate/severe concussion (severity determined on phone screening).
   4. No history of RHI including participation in contact and collision sports (i.e., football, ice hockey, rugby, soccer, lacrosse, wrestling, boxing gymnastics, martial arts, kickboxing), or military service (refers to active combat experience or combat training involving exposure to IED blasts or combatant stick training). These are examples and there might be instances of other RHI sources that could be exclusionary as determined by investigators.
   5. BMI of 24 or higher to be similar in body habitus to former professional and college football players.
   6. Must have at least 2 years of post-secondary education at a 4-year accredited college or university or have an associate's degree if they did not attend a 4-year accredited college or university.
3. AD-CI (n=50) will come from the local ADRCs where Clinical Dementia Rating (CDR) and amyloid biomarker status are known for most participants being followed annually. Inclusion criteria include:

   1. CDR of 0.5-1.0
   2. Positive amyloid PET or CSF AD biomarker within 12 months of study visit (done as part of their participation in the local ADRCs and/or clinical care).
   3. No history of RHI including participation in contact and collision sports (i.e., football, ice hockey, rugby, soccer, lacrosse, wrestling, boxing gymnastics, martial arts, kickboxing), or military service (refers to active combat experience or combat training involving exposure to IED blasts or combatant stick training). These are examples and there might be instances of other RHI sources that could be exclusionary as determined by investigators.
   4. BMI of 24 or higher to be similar in body habitus to former professional and college football players.
   5. No prior anti-amyloid monoclonal antibody treatments or therapeutic trials targeting amyloid or tau prior to initiating study
4. Tracer comparison sub-sample: 20 professional football players from DIAGNOSE-I will have FTP and MK-6240 tau PET (done at the same site, scanner). The 20 participants at highest risk for having CTE pathology will be selected based on the following:

   1. 60+ years old to increase likelihood of meaningful pathology
   2. Must have played professionally
   3. Must have dementia as defined by a CDR of 1.0
   4. Participant was amyloid PET negative at the baseline DIAGNOSE-I evaluation to rule out potential confounding from AD

For newly recruited, those individuals who meet any of the following criteria are not eligible for enrollment as study participants.

Exclusion Criteria:

1. Unstable medical conditions that confound our ability to diagnose neurodegenerative disease accurately (e.g., active cancer with recent chemotherapy or radiation treatments, unstable heart disease particularly if oxygen dependent, kidney disease requiring dialysis)
2. Neurological conditions that confound our ability to diagnose neurodegenerative disease accurately (e.g., acute clinical stroke, severe traumatic brain injury with ongoing symptoms [post-football for football players])
3. Serious mental Illnesses that confound our ability to diagnose neurodegenerative disease accurately (e.g., active psychosis)
4. Inability to fulfill research protocol requirements due to physical, visual, or hearing impairment
5. English is not primary language
6. Unable to travel to 1 of the five study sites to participate
7. Lack of an adequate informant to be available in-person or by telephone for each annual research evaluation. Informant must be 18 years or older, speaks/visits with the participant at least 1X per week for a minimum of 6 months, agree to complete questionnaires about participant, able to travel to study visit if determined it is needed, and is knowledgeable regarding changes to the participant's cognition, mood and behavior
8. Lack of capacity to provide informed consent (IC) or does not have a legal authorized representative or guardian who can provide surrogate IC
9. Unwilling to attempt to have an MRI
10. If willing to complete MRI, contraindications to 3T MRI (e.g., pacemaker, select aneurismal clip, artificial heart valve, select ear implants, select stents incompatible with 3T MRI, metal fragments or foreign objects in the eyes, skin or body, etc.)

For all participants (retention and expansion), the following will be exclusionary for participating in PET scan activities:

1. Medical radiation exposure will be assessed by the study physician. If the candidate participant has had more than one research nuclear medicine study in the prior 12 months, study inclusion will require joint PI approval.
2. Investigational agents are prohibited 30 days prior to entry
3. Initiated medication (investigational or for clinical care) against tau or amyloid proteins prior to their baseline study visit
4. History of a relevant severe drug allergy or hypersensitivity
5. Inability to urinate
6. Any serious illness that, in the study physician's opinion could interfere with the completion of the PET scans or post a potential safety risk

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Former National Football League Players, Former Varsity Level College Football Players, Healthy Controls, Alzheimer's Disease with cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Delayed recall memory | 12 months
  Memory will be assessed by the Rey Auditory Verbal Learning Test Delay Recall. The range of scores on this domain is 0 - 15, with a lower score indicating more problems with memory and a higher risk of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alosco, PhD, Principal Investigator — Boston University Alzheimer's Disease and CTE Center
Locations (5):
- United States (5):
  - Banner Alzheimer's Institute (BAI) and Mayo Clinic Arizona, Phoenix, Arizona
  - University of California, San Francisco (UCSF) Alzheimer Disease Research Center (ADRC), San Francisco, California
  - 1Florida ADRC, University of Florida, Gainesville, Florida
  - Boston University Alzheimer Disease Research Center (ADRC), Boston, Massachusetts
  - South Texas ADRC University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No